CLINICAL TRIAL: NCT02945020
Title: A Phase 1, Open-label, Sequential Study to Investigate the Pharmacokinetic Interaction Between Odalasvir, Given as a Single Agent or in Combination With Simeprevir, and Dabigatran Etexilate Mesylate in Healthy Subjects
Brief Title: A Pharmacokinetic Interaction Study Between Odalasvir, Given as a Single Agent or in Combination With Simeprevir, and Dabigatran Etexilate Mesylate in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR108164; 64294178HPC1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; odalasvir; Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Dabigatran etexilate mesylate+Odalasvir+Simeprevir (Experimental): All participants will receive study medications in a fixed sequential order as: a single dose of dabigatran etexilate mesylate 75 milligram (mg) on Days 1, 17 and 26; Odalasvir (ODV) 25 mg once daily from Day 4 to 28; Simeprevir (SMV) 75 mg once daily from Day 20 to 28. The study drugs will be taken orally.
  Interventions: Drug: Dabigatran etexilate mesylate; Drug: Odalasvir (ODV); Drug: Simeprevir (SMV)

INTERVENTIONS:
Drug: Dabigatran etexilate mesylate — Participants will receive dabigatran etexilate mesylate 75 mg, orally.
Drug: Odalasvir (ODV) — Participants will receive ODV 25 mg, orally.
Drug: Simeprevir (SMV) — Participants will receive SMV 75 mg, orally.

SUMMARY:
The purpose of this study is to evaluate the effect of steady-state concentrations of odalasvir (ODV), as a single agent or in combination with simeprevir (SMV), on the single-dose pharmacokinetics of dabigatran etexilate in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a body mass index (BMI: weight in kilogram [kg] divided by the square of height in meters) of 18.0 to 32.0 kilogram per square meter (kg/m^2), extremes included, and a body weight not less than 50.0 kg
* Participant must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. If there are abnormalities, the participant may be included only if the Investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the Investigator
* Participant must have a blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeters of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic. If blood pressure is out of range, up to 2 repeated assessments are permitted
* Female participant, except if postmenopausal, must have a negative highly sensitive serum beta human chorionic gonadotropin at screening
* Participant must be non-smoker for at least 6 months prior to the first study drug administration

Exclusion Criteria:

* Participant has a history of liver or renal insufficiency (estimated creatinine clearance below 90 milliliter per minute (mL/min) calculated using the Cockcroft-Gault formula or below 90 mL/min/1.73 square meter (m^2) for estimated glomerular filtration rate [eGFR] according to the Chronic Kidney Disease Epidemiology Collaboration equation [CKD-EPI]), significant cardiac, vascular, pulmonary, gastrointestinal (such as significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability), endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances
* Participant has any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the particiapant (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Participant with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticaria
* Participant has known allergies, hypersensitivity, or intolerance to odalasvir (ODV), simeprevir (SMV) or dabigatran etexilate mesylate or their excipients
* Participant has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at screening

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2017-01-09 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Analyte Concentration (Cmax) of Dabigatran | Day 1, 17 and 26 (predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16, 24, 48, and 72 hours post dose)
  Cmax is the maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) of Dabigatran | Day 1, 17 and 26 (predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16, 24, 48, and 72 hours post dose)
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Dabigatran | Day 1, 17 and 26 (predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16, 24, 48, and 72 hours post dose)
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(last)/lambda(z); wherein AUC(0-last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Baseline, up to follow-up (Approximately 43 days)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Tempe, Arizona, United States